CLINICAL TRIAL: NCT04912141
Title: Conestat Alfa (a Recombinant Human C1 Esterase Inhibitor) for the Prevention of Acute Kidney Injury After Non-ST Elevation Myocardial Infarction: a Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 2, Dose-finding Study
Brief Title: Prevention of Acute Kidney Injury in Patients With NSTEMI
Acronym: AKI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lower than expected study enrolment rate. New strategic considerations.
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C1 5201
Record Dates: First submitted 2021-05-21; First posted 2021-06-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-12

CONDITIONS: Non-ST Elevation Myocardial Infarction (NSTEMI)
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — conestat alfa

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter, phase 2, dose-finding.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conestat alfa 50 U/kg - Placebo (Placebo Comparator): 50 U/kg conestat alfa pre-angiography and placebo 3 hours after the first dose
  Interventions: Drug: conestat alfa or placebo
- Conestat alfa 50 U/kg - Conestat alfa 50 U/kg (Active Comparator): 50 U/kg conestat alfa pre-angiography and 3 hours after the first dose
  Interventions: Drug: conestat alfa or placebo
- Conestat alfa 100 U/kg - Conestat alfa 50 U/kg (Active Comparator): 100 U/kg conestat alfa pre-angiography and 50 U/kg conestat alfa 3 hours after the first dose
  Interventions: Drug: conestat alfa or placebo
- Placebo - Placebo (Placebo Comparator): Placebo pre-angiography and 3 hours after the first dose
  Interventions: Drug: conestat alfa or placebo

INTERVENTIONS:
Drug: conestat alfa or placebo — Conestat alfa will be dosed by body weight at 50 U/kg (maximum 4200 U) or 100 U/kg (maximum 8400 U).
  Placebo will consist of normal saline (NaCl 0.9%). The interventions will be given to the patients by IV-line.
  Other Names: Ruconest

SUMMARY:
A randomized, double-blind, placebo-controlled, multi-center, phase 2 clinical study in patients with NSTEMI undergoing urgent coronary angiography. Approximately 220 patients with CKD and acute NSTEMI, who are scheduled for an urgent coronary angiography (within 72 hours after admission and/or diagnosis of NSTEMI).

DETAILED DESCRIPTION:
Approximately 220 patients with chronic kidney disease (CKD) and acute NSTEMI, who are scheduled for an urgent coronary angiography (within 72 hours after admission and/or diagnosis of NSTEMI) will be screened for the study. Only patients with acute NSTEMI presumed to be a spontaneous myocardial infarction, related to atherosclerotic plaque rupture, ulceration, fissuring, erosion, or dissection (i.e. type 1) are eligible. Written informed consent will be obtained before urgent coronary angiography. Patients with NSTEMI will typically undergo coronary angiography within 72 hours after admission and/or diagnosis of NSTEMI. It is estimated that 70% of these patients will have PCI. Randomization will continue until the 160th patient has had a PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by a signature and date of the patient
2. Age 18-85 years
3. Acute NSTEMI as anticipated to be type 1 (expert opinion by the cardiologist before coronary angiography) and scheduled for urgent coronary angiography
4. Documented kidney disease existing for ≥3 months OR Two estimated glomerular filtration rate (eGFR) measurements of <60ml/min/1.73m2 as calculated by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) study equation and at least 6 hours apart OR eGFR of <50 mL/min//1.73m2 as calculated by using the CKD-EPI study equation at presentation
5. At least one of the following risk factors for AKI: diabetes mellitus, age >60 years, established cardiovascular disease, heart failure with reduced ejection fraction, anemia

Exclusion Criteria:

1. Contraindications to the class of drugs under study (C1 esterase inhibitors), e.g. known hypersensitivity or allergy to class of drugs or the IMP
2. History or suspicion of allergy to rabbits
3. Women who are pregnant or breast feeding
4. ST elevation myocardial infarction or unstable angina
5. Cardiogenic shock requiring mechanical support
6. Non-cardiac comorbidity with expected survival <6 months
7. Acute urinary tract infection (e.g. cystitis, pyelonephritis).
8. Liver cirrhosis (any Child-Pugh score)
9. Dialysis or eGFR <20 and >59mL/min/1.73 m2 at baseline (d0)
10. Incapacity or inability to provide informed consent
11. Participation in another study with investigational drug within 30 days preceding, and during the present study
12. Previous enrolment into the current study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Urinary NGAL | 24 hours after PCI
  Evaluation of the peak change of urinary NGAL, an established biomarker of AKI, within 24 hours after PCI

SECONDARY OUTCOMES:
Urinary NGAL | within 24 hours after angiography
  The peak change of urinary NGAL within 24 hours after angiography for the total group including PCI and non-PCI patients
Serum creatinine | within 72 hours after angiography
  The incidence of acute kidney injury (AKI) as defined by a serum creatinine change of ≥26.5 µmol/L or a serum creatinine change of ≥1.5 times baseline within 72 hours after angiography.
Serum cystatin C | 24 hours after angiography
  The incidence of a serum cystatin C change of ≥10% 24 hours after angiography.
Troponin T | within 72 hours after angiography
  The change of troponin T within 72 hours (area under the curve, AUC0-72) after angiography
Troponin T | measured once at 72 hours after angiography
  The peak change of troponin
Creatine kinase | measured once at 72 hours after angiography
  The peak change of creatine kinase
N-terminal pro-brain natriuretic peptide | at 72 hours after angiography
  N-terminal pro-brain natriuretic peptide (NT-proBNP) measured once at 72 hours after angiography

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Relan, MD, Study Director — Pharming Technologies BV
Locations (4):
- Switzerland (4):
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - University Hospital Geneva, Geneva
  - Fondazione Istituto Cardiocentro Ticino, Lugano

IPD SHARING:
Plan to Share IPD: No